CLINICAL TRIAL: NCT05408793
Title: Evaluating the Efficacy of Transcranial Pulse Stimulation (TPS) on Individuals with Autism Spectrum Disorder (ASD)- a Double-blinded, Randomized, Sham-controlled Trial
Brief Title: Effects of Transcranial Pulse Stimulation on ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPU_HSEARS20220228005
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; High-functioning Autism
Keywords: efficacy and safety; transcranial pulse stimulation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, sham-controlled trial.
Who Masked: Participant, Investigator
Masking Description: Double-blind. Participants and interventionists will be blinded to the random allocation to either the verum TPS group or the sham TPS group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Pulse Stimulation (TPS group) (Experimental): Subjects in the TPS group will be given 6 verum TPS sessions (Pulse: 800 / session) across two weeks time, with 3 sessions per week.
  Interventions: Device: Transcranial Pulse Stimulation
- Sham TPS Group (Sham Comparator): Subjects in the Sham TPS group will be given 6 sham TPS sessions across two weeks time, with 3 sessions per week.
  Interventions: Device: Transcranial Pulse Stimulation

INTERVENTIONS:
Device: Transcranial Pulse Stimulation — A total of 36 participants (both TPS group and the sham-control group) will receive six 30 minute-TPS sessions (800 pulse in each session, total: 4800 pulse) in 2 weeks' time (i.e., 3 sessions (Monday, Wednesday, Friday) per week, total: 3 hours), on a 1: 1 allocation ratio. Participants will be followed up immediately after the post-stimulation and at 1-month and 3-month period after the intervention. A 2-week TPS intervention alongside with 3-month follow-up is sufficient enough to test the effects of TPS on autism symptoms.

SUMMARY:
The aim of this study is to evaluate the efficacy and tolerability of TPS on young adolescents with ASD. Methods: This is a two-armed, randomized, double-blinded, sham-controlled trial. Sampling: A total number of 36 subjects, aged between 12 to 17, diagnosed with ASD, will be recruited. Individuals with a Childhood of Autism Rating Scale (CARS) score ≤ 30 (i.e., no ASD) will be excluded. Recruitment: Subjects will be recruited from the community. Block randomization will be performed to allocate subjects to either the verum TPS group or the sham TPS group on a 1: 1 ratio. Interventionists and subjects will be blinded in the randomization process. Intervention: Intervention: Six 30-minures TPS sessions will be delivered to the verum TPS group (800 pulse in each session, total: 4800 pulse) in consecutive two weeks. The treatment brain region is targeted at the right temporoparietal junction (rTPJ). The sham- controlled group will be given 6 sham TPS sessions. Data collection: All participants are required to undertake pre-and-post fMRI and resting-MRI before the TPS procedures. Outcomes: Primary outcome of this study is CARS, and secondary outcomes include Autism Spectrum Quotient (AQ), Australian scale for Asperger's syndrome (ASAS), Social Responsive Scale (SRS), Faux Pas Recognition Test (FPRT), Stroop test, working memory, Clinical global impression - severity and improvement scale (CGI-S and CGI -I) and neuroimaging. All outcome measures will be assessed at baseline, two weeks immediately after intervention and at 1-month and 3-months follow-up.

DETAILED DESCRIPTION:
Primary objective:

1. Participants in the verum TPS group will have a significant reduction in CARS score at posttreatment compared with the sham TPS group.

   Secondary objectives:
2. Participants in the verum TPS group will have significant improvement in Autism Spectrum Quotient (AQ), compared with the sham TPS group.
3. Participants in the verum TPS group will have significant improvement in the Social Responsiveness Scale (SRS), compared with the sham TPS group.
4. Participants in the verum TPS group will have significant improvement in Faux Pas Recognition Test, compared with the sham TPS group.
5. Participants in the verum TPS group will have significant improvement in Stroop test, compared with the sham TPS group.
6. Participants in the verum TPS group will have significant improvement in Clinical global impression - severity and improvement scale (CGI-S and CGI -I) compared with the sham TPS group.
7. Participants in the verum TPS group will have significant brain function connectivity at posttreatment fMRI and resting-state MRI compared to the sham TPS group.

Sample size Based on an RCT with similar design, the estimated effect size of rTMS is 0.5. By adapting an ANOVA 2x2 repeated measures with 95% significance and a power of 0.8, a sample size of 36 will be required in total (18 subjects per group).

Research plan and Methodology Methods Trial Design: In this study, the investigators will use a double-blind randomized controlled trial design with two-armed repeated measures. The trial design complies with the Consolidated Standards of Reporting Trials (CONSORT) statement. In this two-armed design, investigators will use TPS as an intervention group and a waitlist control group. A sham-control group is appropriate for comparing the effect of the TPS on the intervention group to that of those not receiving the TPS treatment at the same timepoints Both groups will be measured at baseline (T1), immediately after the intervention (T2), at the 1-month (T3) and 3-month follow-up (T4). Based on the previous studies, a 3-month follow-up is sufficient to assess the long-term sustainability of the TPS intervention.

Intervention (Transcranial Pulse Stimulation) Purpose of the intervention: The key tenets of the TPS intervention is neuromodulation, i.e., using ultrasound-based brain stimulation techniques to modulate the human brain in a focal and targeted manner. Intervention dose: Each participant should have the pre-treatment MRI scan performed in the University Research Facility in Behavioural and Systems Neuroscience, PolyU prior coming to the first intervention session. All participants (both TPS group and the sham-control group) will receive six 30 minute-TPS sessions (800 pulse in each session, total: 4800 pulse) in 2 weeks' time. Participants will be followed up immediately after post-stimulation in Week 2, and at 1-month and 3- month period after the intervention. The investigators believe that a 2-week TPS intervention is sufficient enough to test the effects of TPS on autism symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 12 -17 years of age
2. Chinese ethnicity
3. Diagnosis of Autistic Spectrum Disorder that meets the criteria of the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
4. No change in their management including medications or non-pharmacological intervention
5. Currently taking prescribed psychotropic medications for ≥ 3 months

Exclusion Criteria:

1. A DSM-5 diagnosis other than ASD
2. Concomitant major medical or neurological conditions, such as significant global developmental delay, skull defect, abnormal mass or tumor, or epilepsy
3. A CARS score ≤ 30 (i.e., no ASD)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Autism severity | Changes in CARS scores from baseline at 3 months
  The Childhood Autism Rating Scale (CARS) is a 15-item behavioral rating scale developed to identify autism and examine its severity. Total scores range from a low of 15 to a high of 60; scores below 30 indicate that the individual is in the non-autistic range, scores between 30 and 36.5 indicate mild to moderate autism, and scores from 37 to 60 indicate severe autism.

SECONDARY OUTCOMES:
Autistic traits | Changes in AQ scores from baseline at 3 months
  Autism Spectrum Quotient (AQ) - adolescent version is a quick and quantitative self-report instrument for assessing how many autistic traits any adult has. The minimum score on the AQ is 0 and the maximum 50.
Social deficits | Changes in SRS from baseline at 3 months
  The Social Responsiveness Scale (SRS) is an instrument measuring the continuum of autism symptom severity which is commonly used in children and adolescents between the ages of 4 and 18 years. Parents rate on each item on a 4-item Likert scale (0-4). The higher the scores, the more severe the social deficits.
Asperger's Syndrome | Changes in ASAS from baseline at 3 months
  Australian scale for Asperger's syndrome (ASAS) is a scale used to screen the behaviours and abilities indicative of Asperger's Syndrome in subjects older than 6 years old. It has 25 item and can be rated by parents/teachers/professionals who know the child.
Theory of Mind and Social Cognition | Changes in FPRT from baseline at 3 months
  Faux Pas Recognition Test (FPRT) is a very common advanced test to measure the theory of mind and social cognition
Executive Function | Changes in Stroop test from baseline at 3 months
  Stroop test is commonly used to assess the inhibition control component of executive function. It is testing the subject's ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute.
Working memory | Changes in WMTB from baseline at 3 months
  Working Memory Test Battery (WMTB), which includes two verbal storage-only tasks (i.e. digital recall and word list recall), two complex memory span tasks (i.e. backward digit recall and counting recall), and two visuospatial storage tasks (block recall and variant- visual-pattern test).
Clinical Global Impression | Changes in WMTB from baseline at 3 months
  CGI-S is a 7-point clinician rating scale is based upon observed and reported symptoms, behaviour, and function in the past seven days. CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Neuroimaging | MRI will be assessed at baseline at immediately and 2 weeks after post-stimulation
  Participants will receive pre and post treatment MRI scan to measure any changes in structural and functional connectivity changes in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Teris Cheung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing HongKongPolyU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu CL, Matt E, Fong TKH, Lam JYT, Chau B, Cheng CPW, Beisteiner R, Cheung T. Associations Between Brain Network Connectivity and Cognitive Measures in Autism Spectrum Disorder: A Post Hoc Analysis of a Parent Study "Evaluating the Safety and Efficacy of Transcranial Pulse Stimulation on Autism Spectrum Disorder". Autism Res. 2025 Oct;18(10):1965-1977. doi: 10.1002/aur.70093. Epub 2025 Aug 21. PMID 40841688
- [Derived] Cheung T, Ho YS, Fong KH, Lam YTJ, Li MH, Tse AC, Li CT, Cheng CP, Beisteiner R. Evaluating the Safety and Efficacy of Transcranial Pulse Stimulation on Autism Spectrum Disorder: A Double-Blinded, Randomized, Sham-Controlled Trial Protocol. Int J Environ Res Public Health. 2022 Nov 24;19(23):15614. doi: 10.3390/ijerph192315614. PMID 36497688